CLINICAL TRIAL: NCT00003127
Title: Phase II Trial of Paclitaxel and Carboplatin With Amifostine in Advanced Recurrent or Refractory Endometrial Adenocarcinoma
Brief Title: S9720 Combination Chemotherapy in Treating Patients With Metastatic, Recurrent, or Refractory Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065890; SWOG-S9720 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-06-24 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Endometrial Cancer
Keywords: stage IV endometrial carcinoma; recurrent endometrial carcinoma; endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma; endometrial clear cell carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Amifostine; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carbo, taxol, amifostine (Experimental): carbo, taxol, amifostine
  Interventions: Drug: amifostine trihydrate; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: amifostine trihydrate — 740 mg/m2 IV, Day 1, q 28 days X 6 cycles
  Other Names: ethyol
Drug: carboplatin — target AUC=6, IV Day 1, q 28 days X 6 cycles
  Other Names: carbo
Drug: paclitaxel — 175 mg/m2, IV, Day 1 q 28 days X 6 cycles
  Other Names: Taxol

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with metastatic, recurrent, or refractory endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of paclitaxel and carboplatin with amifostine on progression free survival and overall survival in patients with metastatic or recurrent epithelial endometrial carcinoma not amenable to surgery or radiotherapy. II. Evaluate response (confirmed and unconfirmed partial response and complete response) rate to this regimen in this patient population. III. Assess the nature and degree of toxicity of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 3 hours, then amifostine IV over 10 minutes, followed fifteen minutes later by carboplatin IV over 30-60 minutes on day 1. Courses repeat every 28 days. Treatment continues for 6 courses in the absence of disease progression. Patients are followed every 6 months for 2 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 35 to 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic, recurrent, or refractory epithelial endometrial carcinoma Must be one of the following histologic types: Endometrioid adenocarcinoma Villoglandular Secretory Ciliated Endometrioid adenocarcinoma with squamous differentiation Serous carcinoma Clear cell carcinoma Mucinous carcinoma Squamous carcinoma Mixed types of carcinoma Undifferentiated carcinoma Must not be amenable to surgery or radiotherapy Documented evidence of progression at site if the only site of measurable disease has been irradiated Metastatic sites need not be biopsied Measurable disease

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 25 mL/min Other: At least 5 years since other prior malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy No more than 1 prior biologic therapy regimen Chemotherapy: No concurrent chemotherapy No prior taxane for any reason No more than 2 prior chemotherapy courses used for the sole purpose of radiosensitization during primary definitive therapy allowed No other prior chemotherapy Endocrine therapy: No concurrent hormonal therapy Prior hormonal or other endocrine therapy allowed Radiotherapy: No concurrent radiotherapy except to sites of bone metastases for palliative control of pain Prior radiotherapy to no more than 30% of bone marrow allowed At least 4 weeks since radiotherapy and recovered Surgery: Prior surgery allowed Must have recovered from surgery and any complication therefrom

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 1998-02; Primary Completion 2003-04 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 6 months
  from date of registration to date of first observation of progressive disease, deathe due to any cause, or early discontinuation of treatment.

SECONDARY OUTCOMES:
overall survival | 6 months
  From date of registration to date of death due to any cause
response | after 12 and 24 weeks
  Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No disease progression. No new lesions.
toxicity | Weekly X 3, q 4 weeks X 6 cycles
  assessment per SWOG toxicity criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sidney A. Scudder, MD, Study Chair — University of California, Davis
Locations (94):
- United States (94):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Scudder SA, Liu PY, Wilczynski SP, Smith HO, Jiang C, Hallum AV 3rd, Smith GB, Hannigan EV, Markman M, Alberts DS; Southwest Oncology Group. Paclitaxel and carboplatin with amifostine in advanced, recurrent, or refractory endometrial adenocarcinoma: a phase II study of the Southwest Oncology Group. Gynecol Oncol. 2005 Mar;96(3):610-5. doi: 10.1016/j.ygyno.2004.11.024. PMID 15721401
- [Result] Scudder SA, Liu PY, Smith HO, et al.: Paclitaxel (PCT) and carboplatin (C) with amifostine (A) in advanced or recurrent endometrial cancer: a Southwest Oncology Group trial (S9720). [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-819, 2001.